CLINICAL TRIAL: NCT05227846
Title: A Phase 1 Dose Escalation Study of Human Umbilical Cord-derived Mesenchymal Stem Cells for the Treatment of Decompensated Cirrhosis (MSC-DLC-1)
Brief Title: Human Umbilical Cord-derived Mesenchymal Stem Cells for Decompensated Cirrhosis (MSC-DLC-1)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing 302 Hospital (Other)
Collaborators: Vcanbio Cell and Gene Engineering Corp., Ltd. (Industry)
Responsible Party: Principal Investigator, Fu-Sheng Wang, Head of Treatment and Research Center for Infectious Diseases, Principle Investigator, Clinical Professor, Beijing 302 Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSC-DLC-1
Record Dates: First submitted 2022-01-26; First posted 2022-02-07 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Decompensated Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Human Umbilical Cord-derived Mesenchymal Stem Cells (Experimental): Standard of care (SOC) plus a dose-escalation with 4 cohorts with 3-6 subjects/cohort who receive doses of 5, 10，15 and 20 ×10E7 cells. Proceed from lower dose to next higher dose if no safety concerns for each cohort.
  Interventions: Biological: Human Umbilical Cord-derived Mesenchymal Stem Cells

INTERVENTIONS:
Biological: Human Umbilical Cord-derived Mesenchymal Stem Cells — Human Umbilical Cord-derived Mesenchymal Stem Cells will be administered intravenously.

SUMMARY:
This is a Phase 1, open label, dose escalation clinical trial of human umbilical cord-derived mesenchymal stem cells for the treatment of decompensated cirrhosis. The purpose of this study is to assess the safety of human umbilical cord-derived mesenchymal stem cells in patients with decompensated cirrhosis.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the safety of intravenous infusion of human umbilical cord-derived mesenchymal stem cells in patients with decompensated cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to provide written informed consent;
2. Aged 18 to 75 years (including 18 and 75 years), male or female;
3. Patients diagnosed with decompensated liver cirrhosis based on clinical findings, laboratory tests, imaging findings and/or representative pathological findings (decompensated liver cirrhosis is defined as the occurrence of at least one serious complication, including esophageal and gastric varices bleeding, hepatic encephalopathy, ascites, spontaneous bacterial peritonitis and other serious complications);
4. Child-Turcotte-Pugh (CTP) score 7 to 12 points.

Exclusion Criteria:

1. Appearance of active variceal bleeding, overt hepatic encephalopathy (HE), refractory ascites or hepatorenal syndrome within 1 month prior to screening visit.
2. Uncontrolled severe infection within 2 weeks of screening.
3. Hepatitis B virus (HBV) DNA ≥ detection limit at the time of screening.
4. Patients with hepatitis B virus-related decompensated liver cirrhosis may discontinue antiviral therapy during the study, or those who with antiviral therapy for HBV for less than 12 months.
5. Patients with hepatitis C virus-related decompensated liver cirrhosis may discontinue antiviral therapy during the study, or those who with antiviral therapy for HCV for less than 12 months.
6. Patients under treatment with corticosteroids for autoimmune hepatitis for less than 6 months.
7. Trans-jugular intrahepatic portosystemic shunts (TIPS) insertion within 6 months prior to study inclusion.
8. Active drinkers with alcohol-related decompensated cirrhosis are unwilling to stop alcohol abuse after inclusion.
9. Severe jaundice (serum total bilirubin level ≥ 170μmol/L); Significant renal insufficiency (serum creatinine ≥ 1.2 times upper normal limit); Severe electrolyte abnormality (serum sodium level < 125 mmol/L); Severe leukopenia (white blood cell count < 1 × 10E9/L).
10. Patients with biliary obstruction, hepatic vein, portal vein, splenic vein thrombosis and portal vein spongiosis.
11. Patients with surgical history such as splenic cut-off flow and portal body shunt.
12. Patients with confirmed or suspected malignancies.
13. Patients with a prior history of major organ transplantation or complicated with significant disease of heart, lung, kidney, blood, endocrine and other systems.
14. Drug abuse, drug dependence and patients who receive methadone treatment or with psychosis.
15. HIV seropositivity.
16. Those who have received blood transfusion or other blood products within 1 month prior to screening visit.
17. Pregnancy, lactation or with recent fertility plan.
18. Highly allergic or have a history of severe allergies.
19. Participants in other clinical trials within the last 3 months.
20. Any other clinical condition which the investigator considers would make the patient unsuitable for the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events Incidence of Adverse Events | from baseline to 28th day
Change in Model for End-Stage Liver Disease (MELD) score from baseline to 28th day | at 28th day
  The Model for End-stage Liver Disease (MELD) is a scoring system that evaluates the liver function reserve and prognosis of patients with chronic liver disease by creatinine, international normalized ratio (INR), and bilirubin-conjugated cirrhosis etiology.
  The MELD score is calculated by the formula: R = 9.6 × ln (creatinine mg/dl) + 3.8 × ln (bilirubin mg/dl) + 11.2 × ln (INR) + 6.4 × etiology, and the results are taken as integers. ( 0 for cholestatic and alcoholic cirrhosis and 1 for other causes of cirrhosis such as viruses).

SECONDARY OUTCOMES:
Change in Model for End-Stage Liver Disease (MELD) score from baseline to 3 days, 7days, 14 days, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months, 21 months, and 24 months | 3 days, 14 days, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months, 21 months, and 24 months
Incidence of each complication associated with decompensated cirrhosis | up to 24 months
liver transplant-free survival | up to 24 months
Incidence of liver failure | up to 24 months
plasma albumin (ALB) | up to 24 months
plasma prealbumin (PALB) | up to 24 months
total bilirubin (TBIL) | up to 24 months
serum cholinesterase (CHE) | up to 24 months
prothrombin time (PT) | up to 24 months
  Prothrombin time (PT) is a blood test that measures the time it takes for plasma to clot, to check for bleeding problems, or to check whether medicine to prevent blood clots is working.
Child-Turcotte-Pugh (CTP) score | up to 24 months
  Child-Turcotte-Pugh (CTP) score is a scoring system that evaluates the liver function.
  Maximum is 15, minimum is 5. Higher scores mean a worse outcome.
EuroQol Group 5-Dimension Self-Report Questionnaire (EQ-5D) | up to 24 months
  Quality of life assessment. Maximum is 5, minimum is 1. Lower scores mean a better outcome.
Incidence of liver cancer | up to 24 months
ChronicLiver Disease Questionnaire (CLDQ) | up to 24 months
  Quality of life assessment. The Chronic Liver Disease Questionnaire (CLDQ) was developed as an evaluative instrument to measure longitudinal change in health status within individuals with chronic liver disease. In addition to measuring both physical and mental health, the instrument was designed to be a disease-specific tool for assessing areas of function important to patients with chronic liver disease. Maximum is 7, minimum is 1. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Sheng Wang, MD, PhD, Study Chair — Beijing 302 Hospital
Locations (1):
- Beijing 302 Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
After approval from the steering committee and the Human Genetic Resources Administration of China, this trial data can be shared with qualifying researchers who submit a proposal with a valuable research question. A contract should be signed.

REFERENCES:
- [Derived] Shi L, Zhang Z, Mei S, Wang Z, Xu Z, Yao W, Liu L, Yuan M, Pan Y, Zhu K, Liu K, Meng F, Sun J, Liu W, Xie X, Dong T, Huang L, Meng F, Fu JL, Li Y, Zhang C, Fan X, Shi M, Zhang Y, Li Y, Xie WF, Zhang P, Wang FS. Dose-escalation studies of mesenchymal stromal cell therapy for decompensated liver cirrhosis: phase Ia/Ib results and immune modulation insights. Signal Transduct Target Ther. 2025 Jul 29;10(1):238. doi: 10.1038/s41392-025-02318-4. PMID 40721581
- [Derived] Wang Z, Li T, Zhang Z, Yuan M, Shi M, Wang FS, Linghu EQ, Shi L. Human umbilical cord-derived mesenchymal stem cells for the treatment of decompensated cirrhosis (MSC-DLC-1): a dose-escalation, phase I trial protocol. BMJ Open. 2023 Dec 30;13(12):e078362. doi: 10.1136/bmjopen-2023-078362. PMID 38159943